CLINICAL TRIAL: NCT06618469
Title: Effects of Resistance Training Programes At Different Intensities on Musculoskeletal, Metabolic, Lipid, Immunological, Inflammatory, Well-being and Functional Parameters in Older Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Oxidative Pathology Unit of the Department of Biochemistry and Molecular Biology, University of Valencia. (Unknown)
Responsible Party: Principal Investigator, Juan C. Colado, Chaired Full Professor of Physical Education and Sports, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H1395923230221; OTR2015-140931NVES (Other Grant/Funding Number: MAPFRE Fundation)
Record Dates: First submitted 2024-09-18; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Aging
Keywords: Aging; Dose-response; Exercise intensities; Oxidative stress; Physical activity; Bone health; Neuromuscular physiology
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a randomized, duoble-blind (sport scientiest assistance/care assistance-outcome assessor), 6 arms prospective parallel design clinical trial. The older adults will be recruited from the Municipal Activity Centers for Older People located in Valencia and will be randomized in a prospective clinical trial study with a 6 parallel arms study design to a tubes or bands or water resistance training modalities performed at different intensities or a control group over a 32 weeks period.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: For masking the participants, the investigators will not inform participants of what group they will be in. For outcome assessor, data collectors and data analysts independent people will be use, and if this is not possible, a random code will be created for each participant so that it is not possible to identify which group belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Elastic band-based resistance training program at high intensity (HI) (Experimental)
  Interventions: Behavioral: Elastic band-based resistance training program at high intensity (HI)
- Elastic band-based resistance training program at moderate-high intensity (MHI-bands) (Experimental)
  Interventions: Behavioral: Elastic band-based resistance training program at moderate-high intensity (MHI-bands)
- Elastic band-based resistance training program at moderate intensity (MI) (Experimental)
  Interventions: Behavioral: Elastic band-based resistance training program at moderate intensity (MI)
- Elastic tubes-based resistance training program at moderate-high intensity (MHI-tubes) (Experimental)
  Interventions: Behavioral: Elastic tubes-based resistance training program at moderate-high intensity (MHI-tubes)
- Water-based resistance training program at moderate intensity (WMI) (Experimental)
  Interventions: Behavioral: Water-based resistance training program at moderate intensity (WMI)
- Control group (No Intervention): Participants randomized into the CONTROL group will not undertake any formal intervention and will be asked to maintain their usual physical activity habits and diet.

INTERVENTIONS:
Behavioral: Elastic band-based resistance training program at high intensity (HI) — The training session will consist of 5-10 minutes of general warm-up (joint- mobility and aerobic exercises at low intensity); 35-40 minutes of the main part, which comprised six resistance exercises, three for upper limbs (upright rowing, incline rowing, and elbow curl) and three for lower limbs (narrow stance squat, lunge, and standing hip abduction) along with coordination exercises during the active rests; and 5-10 minutes of the cool-down routine (respiratory and flexibility exercises). The participants will perform 6 submaximal repetitions using elastic bands equivalent to 85% of the one-repetition maximum per exercise (high load/intensity training sessions). The perceived exertion level on the OMNI-RES scale progressed from 6-7 to 8-9 . The number of sets per exercise progressed from 3 to 4. The speed of execution of the exercises was controlled using a metronome marking the cadence (2s of concentric and eccentric phase).
  Other Names: 1
  Arms: Elastic band-based resistance training program at high intensity (HI)
Behavioral: Elastic band-based resistance training program at moderate-high intensity (MHI-bands) — The training session will consist of 5-10 minutes of general warm-up (joint- mobility and aerobic exercises at low intensity); 35-40 minutes of the main part, which comprised six resistance exercises, three for upper limbs (upright rowing, incline rowing, and elbow curl) and three for lower limbs (narrow stance squat, lunge, and standing hip abduction) along with coordination exercises during the active rests; and 5-10 minutes of the cool-down routine (respiratory and flexibility exercises). The participants will perform 6 submaximal repetitions using elastic bands equivalent to 75-80% of the one-repetition maximum per exercise (high to moderate load/intensity training sessions). The perceived exertion level on the OMNI-RES scale progressed from 6-7 to 8-9 . The number of sets per exercise progressed from 3 to 4. The speed of execution of the exercises was controlled using a metronome marking the cadence (2s of concentric and eccentric phase).
  Other Names: 2
  Arms: Elastic band-based resistance training program at moderate-high intensity (MHI-bands)
Behavioral: Elastic band-based resistance training program at moderate intensity (MI) — The training session will consist of 5-10 minutes of general warm-up (joint- mobility and aerobic exercises at low intensity); 35-40 minutes of the main part, which comprised six resistance exercises, three for upper limbs (upright rowing, incline rowing, and elbow curl) and three for lower limbs (narrow stance squat, lunge, and standing hip abduction) along with coordination exercises during the active rests; and 5-10 minutes of the cool-down routine (respiratory and flexibility exercises). The participants will perform 6 submaximal repetitions using elastic bands equivalent to 65-70% of the one-repetition maximum per exercise (moderate load/intensity training sessions). The perceived exertion level on the OMNI-RES scale progressed from 6-7 to 8-9. The number of sets per exercise progressed from 3 to 4. The speed of execution of the exercises was controlled using a metronome marking the cadence (2s of concentric and eccentric phase).
  Other Names: 3
  Arms: Elastic band-based resistance training program at moderate intensity (MI)
Behavioral: Elastic tubes-based resistance training program at moderate-high intensity (MHI-tubes) — The training session will consist of 5-10 minutes of general warm-up (joint- mobility and aerobic exercises at low intensity); 35-40 minutes of the main part, which comprised six resistance exercises, three for upper limbs (upright rowing, incline rowing, and elbow curl) and three for lower limbs (narrow stance squat, lunge, and standing hip abduction) along with coordination exercises during the active rests; and 5-10 minutes of the cool-down routine (respiratory and flexibility exercises). The participants will perform 6 submaximal repetitions using elastic tubes equivalent to 75-80% of the one-repetition maximum per exercise (high to moderate load/intensity training sessions). The perceived exertion level on the OMNI-RES scale progressed from 6-7 to 8-9 . The number of sets per exercise progressed from 3 to 4. The speed of execution of the exercises was controlled using a metronome marking the cadence (2s of concentric and eccentric phase)
  Other Names: 4
  Arms: Elastic tubes-based resistance training program at moderate-high intensity (MHI-tubes)
Behavioral: Water-based resistance training program at moderate intensity (WMI) — The training session will consist of 5-10 minutes of general warm-up (joint- mobility and aerobic exercises at low intensity); 35-40 minutes of the main part, which comprised six resistance exercises, three for upper limbs (upright rowing, incline rowing, and elbow curl) and three for lower limbs (narrow stance leg extension and flexion, hip flexion and extension, and standing hip abduction) along with coordination exercises during the active rests; and 5-10 minutes of the cool-down routine (respiratory and flexibility exercises). The participants will perform in the poll the concentric and eccentric movements of each exercise at maximal velocity during 40 seconds (equivalent to working around 10 repetitions /75% 1RM each exercise). The perceived exertion level on the OMNI-RES scale progressed from 6-7 to 8-9. The number of sets per exercise progressed from 3 to 4.
  Other Names: 5
  Arms: Water-based resistance training program at moderate intensity (WMI)

SUMMARY:
The aging of the global population is recognized by the World Health Organization (WHO) as a major issue due to the disabilities and comorbidities related to this process, with women being the gender most affected. Due to the physiological and psychological age associated declines, physical activity and exercise are proven strategies for reducing the impact of aging. However, it is still unknown what kind of training program could be the most effective in reversing deleterious age-related changes in older adults. Regarding this, the type of training intensity and exercise modality are two key training parameters in exercise programming, and, therefore, different adaptations could be induced in older adults through the modification of these parameters. Furthermore, the type of training device is a significant factor and can act as a barrier or facilitator in older adults' participation in physical activities and exercise programs. Therefore, the research project primary goals are to compare the effects of resistance training programes performed at different intensities and materials during 32 weeks on a variety of physiological parameters in older adults.

DETAILED DESCRIPTION:
This is a randomized clinical trial (RCT) with 6 parallel arms. The subjects will be divided in 6 groups with a randomized technique assigned to a 32-week of: a) progressive elastic band-based resistance training program at high intensity (HI); b) progressive elastic band-based resistance training program at moderate-high intensity (MHI-bands); c) progressive elastic band-based resistance training program at moderate intensity (MI); d) progressive elastic tubes-based resistance training program at moderate-high intensity (MHI-tubes); e) progressive water-resistance training program at moderate intensity (WMI); f) self-management control group (CG). The subjects will be submitted to a 2-session familiarization period and then a 32-week of training program will be performed twice a week.

The exercise groups engaged in progressive elastic-based (bands of tubes) resistance training twice a week with three to four sets of six (HI), 10 (MHI) or 15 (MI) submaximal repetitions including six overall body exercises at a rate of perceived exertion (RPE) of 6-7 in the first four weeks and 8-9 in the remaining weeks on the OMNI-Resistance Exercise Scale (RES). The water-resistance group will perform similar exercises adapted to the water environment at maximal effort (maximal speed in the concentric and eccentric phases of each repetition) during 40 seconds. Members of the control group were instructed to continue their everyday lives.

Oxidative stress, bone health, body composition, neuromuscular strength, physical function, quality of life, lipidic, immune and cardiometabolic profile will be assessed. Oxidative stress status will be assessed in deoxyribonucleic acid (DNA) (urinary 8-oxo-2-deoxyguanosine [8-oxo-dG], lipids (F2-isoprostanes[8-iso-P]; malonaldehyde [MDA], and proteins (protein carbonyls) products together with antioxidant enzymes (superoxide dismutase [SOD] and glutathione peroxidase [GPx]), and thiol redox state (reduced glutathione [GSH], oxidized glutathione [GSSG], and the GSSG/GSH ratio. Bone health will be integrated by measures of areal bone mineral density (aBMD) and the T-score of the lumbar spine (L1-L4 segments, L2-L4 segments, and L1, L2, L3, and L4 individual vertebrae) and proximal femur (femoral neck, trochanter, intertrochanter, Ward's triangle, and total hip in both projects) will be assessed by dual-energy X-ray absorptiometry (DXA). Additionally bone health will be also composed by fracture risk (the 10-year probability of a major osteoporotic fracture and the 10-year probability of a hip fracture), bone turnover markers (BTMs) of bone formation (procollagen type I N propeptide [P1NP], a bone-specific isoform of alkaline phosphatase [bALP]) and bone resorption (a β-isomerized form of C-terminal telopeptide of type I collagen [β-CTx]), and their relationship (bALP/ β-CTx ratio). Body composition (total body mass, total fat mass, total fat-free mass, and total body fat percentage) will be measured by DXA. Moreover, the neuromuscular strength of upper limbs (elbow flexor and extensor muscles) and lower limbs (hip abductor and hip adductor along with knee flexor and extensor muscles) will be assessed through isokinetic dynamometry at low (60°/s) and high (180°/s) velocities. Finally, physical performance will be measured using various functional tests and batteries widely used in the literature, such as the 30 seconds chair stand (30sec-CS) and 30 seconds arm curl (30sec-AC) for muscle strength/endurance of the lower and upper limbs; time up and go (TUG) for dynamic balance/agility; the six-minute walking test (6MWT) for aerobic endurance; five sit-to stand.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* Physically independent (able to walk 100 m without a walking aid and climb 10 steps without rest)
* On the registration waiting list for physical activity at their respective Municipal Activity Centers for Older People (MACOP).
* Sedentary lifestyle (less than one hour of physical activity or exercise a week during the previous six months).
* Medical certificate of suitability or fitness to practice resistance training activities.
* No plans to leave the area during the intervention.
* Cognitive ability to understand and follow the instructions and sign the informed consent form.
* Free of any antioxidant supplements for at least six weeks before the start of this study.

Exclusion Criteria:

* Presence of cardiovascular, musculoskeletal, renal, liver, pulmonary, or neuromuscular and neurological disorders that would prevent the participant from performing the exercises.
* Current or prior (past six months) use of hormone replacement therapy.
* Body weight changes > 10% in the previous year.
* Intake of prescription medications or supplements (e.g., vitamins C, E) that were expected to alter the results of the study (ergogenic, dietary aids, estrogen, beta-blockers, steroid hormones, calcitonin, corticosteroids, glucocorticoids, thiazide diuretics, anticonvulsants, bisphosphonates, raloxifene).
* A history of malignant neoplasms.
* Terminal illness with life expectancy of less than one year.
* Engagement in regular strength training (more than once a week) during the previous six months.
* Participation in another research project (within the last six months) involving dietary, exercise, and/or pharmaceutical intervention.
* Mini mental State Examination lower than 23/30.
* Severe visual or hearing impairment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in DNA oxidative stress | Baseline and 16 weeks
  The oxidative stress of DNA will be assessed via urine collections of 8-oxo-7,8- dihydro-20-deoxyguanosine (8-OHdG) in nmol/mmol creatinine.
Change in lipid peroxidation | Baseline and 16 weeks
  The lipid peroxidation will be assessed via urine and blood collections of 8-isoprostane(nmol /mmol creatinine) and Malondialdehyde (μmol/L)
Change in protein oxidation | Baseline and 16 weeks
  The protein oxidation will be assessed via blood collections of protein carbonyl (nmol/L)
Change in antioxidants enzymes-Superoxid dismutase | Baseline and 16 weeks
  The antioxidants enzymes will be assessed via blood collections of superoxid dismutase (U · mL-1)
Change in antioxidants enzymes-reduced glutathione | Baseline and 16 weeks
  The antioxidants enzymes will be assessed via blood collections of reduced glutathione (nmol/mg protein)
Change in antioxidants enzymes- Glutathione peroxidase | Baseline and 16 weeks
  The antioxidants enzymes will be assessed via blood collections of glutathione peroxidase (IU/g Hb).
Change in antioxidants enzymes-oxidized glutathione | Baseline and 16 weeks
  The antioxidants enzymes will be assessed via blood collections of oxidized glutathione (nmol/mg protein).
Change in antioxidants enzymes-Catalase | Baseline and 16 weeks
  The antioxidants enzymes will be assessed via blood collections of catalase (IU/g Hb).

SECONDARY OUTCOMES:
Change in inflammatory profile | Baseline, 16 and 32 weeks
  The C-reactive protein (mg/L) and interleukin 6 (IL-6) will be assessed via blood collections.
Change in renal and hepatic profile | Baseline, 16 and 32 weeks
  Glutamic-pyruvic transaminase (GPT), glutamic-oxaloacetic transaminase (GOT); gamma-glutamyl transpeptidase (GCT) and alkaline phosphatase (ALP) will be measured.
Change in metabolic profile-glycosylated hemoglobin A1C | Baseline, 16 and 32 weeks
  The metabolic profile will be assessed via blood collections of glycosylated hemoglobin A1C (%).
Change in metabolic profile-basal glucose | Baseline, 16 and 32weeks
  The metabolic profile will be assessed via blood collections of basal glucose (mmol/l).
Change in immune profile-Platelet counts | Baseline, 16 and 32 weeks
  The immune profile will be assessed via blood collections of platelet counts (10*9/L).
Change in immune profile-plateletcrit | Baseline, 16 and 32 weeks
  The immune profile will be assessed via blood collections of plateletcrit (%)
Change in immune profile-mean platelet volum | Baseline, 16 and 32 weeks
  The immune profile will be assessed via blood collections of mean platelet volum (fl).
Change in immune profile-platelet distribution width | Baseline, 16 and 32 weeks
  The immune profile will be assessed via blood collections of platelet distribution width (%).
Change in immune profile-leukocites | Baseline, 16 and 32 weeks
  The immune profile will be assessed via blood collections of platelet counts leukocytes (% and 10*9/L).
Change in immune profile- neutrophils | Baseline, 16 and 32 weeks
  The immune profile will be assessed via blood collections of neutrophils (% and 10*9/L).
Change in immune profile-lymphocytes | Baseline, 16 and 32 weeks
  The immune profile will be assessed via blood collections of lymphocytes (% and 10*9/L).
Change in immune profile-monocytes | Baseline, 16 and 32 weeks
  The immune profile will be assessed via blood collections of monocytes (% and 10*9/L).
Change in immune profile-eosinophils | Baseline, 16 and 32 weeks
  The immune profile will be assessed via blood collections of eosinophils (% and 10*9/L).
Change in immune profile-basophils | Baseline, 16 and 32 weeks
  The immune profile will be assessed via blood collections of basophils (% and 10*9/L).
Change in lipid profile-total cholesterol | Baseline, 16 and 32 weeks
  The lipid profile will be assessed via blood collections: total cholesterol (mg/dL)
Change in lipid profile-high-density lipoprotein cholesterol | Baseline, 16 and 32 weeks
  The lipid profile will be assessed via blood collections: high-density lipoprotein cholesterol (mg/dL).
Change in lipid profile-low-density lipoprotein cholesterol | Baseline, 16 and 32 weeks
  The lipid profile will be assessed via blood collections: low-density lipoprotein cholesterol (mg/dL)
Change in lipid profile-triglycerides | Baseline, 16 and 32 weeks
  The lipid profile will be assessed via blood collections triglycerides (mg/dL)
Change in lipid profile-apolipoprotein B/apolipoprotein A | Baseline, 16 and 32 weeks
  The lipid profile will be assessed via blood collections: apolipoprotein B/apolipoprotein A (ApoB/ApoA) ratio
Change in bone metabolism - Type I procollagen N-terminal propeptide (Bone formation) | Baseline, 16 and 32 weeks
  The bone metabolism will be assessed via blood collections of Type I procollagen N-terminal propeptide (P1NP).
Change in bone metabolism - Bone alkaline phosphatase (Bone formation) | Baseline, 16 and 32 weeks
  The bone metabolism will be assessed via blood collections of bone alkaline phosphatase which are markers marker of bone formation.
Change in bone metabolism - terminal telopeptide of collagen type I (bone resorption) | Baseline, 16 and 32 weeks
  The bone metabolism will be assessed via blood collections of terminal telopeptide of collagen type I (β-CTX- 1) which is a marker of bone resorption.

OTHER OUTCOMES:
Change in isokinetic muscle strength | Baseline, 16 and 32 weeks
  The dynamic maximal concentric muscle strength of the dominant side of hip (flexo-extension and abduction and adduction muscle groups), knee and elbow (flexion and extension muscle groups) and shoulder (flexo-extension) will be measured with an isokinetic dynamometer (Biodex System 4 Pro; Biodex, Shirley, NY) at two angular velocities, 60°/s and 180°/s. Maximal voluntary concentric isokinetic torque will be assessed in Newton-meters (N-m).
Change in maximal muscle hand grip strength | Baseline, 16 and 32 weeks
  The isometric maximal muscle hand grip strength of both hands will be measured with a dynamometer.
Change in maximal isometric strength | Baseline, 16 and 32 weeks
  Maximal isometric strength of upper limbs (seated row exercise), lower limbs (leg press exercise) and back muscles (back extension)
Change in functional performance | Baseline, 16 and 32 weeks
  The functional performance will be assessed with Senior Fitness tests that involve 6 tests: Arm Curl (number of biceps curl in 30 seconds); Chair Stand (stand up from a chair as often as possible within 30s); Back Scratch (for shoulder flexibility, cm between fingertips in the back); Chair sit and reach (for lower flexibility, cm between the extended middle fingers and the tip of the shoe); Up-and-Go (for dynamic balance, time for got up from the chair, walk as quickly as possible around a cone placed 2.4 m from the chair, and resume the seated position); Six-Minute walking test (for aerobic capacity, distance walked in 6 minutes).
Height | Baseline, 16 and 32 weeks
  Height will be recorded to the nearest 0.01 cm using a stadiometer (Seca 711, Hamburg, Germany)
Change in bone mineral density (BMD) | Baseline, 16 and 32 weeks
  BMD (g/cm2) will be assessed for whole body, proximal femur on the non-dominant side (femoral nech, trochanter, intertrochanter, Ward's triangle and total hip) and lumbar spine segments (L1-L4) (L2-L4) (L1-L3) and single vertebrae (L1, L2, L3, L4) will be assessed using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change bone mineral content (BMC) | Baseline, 16 and 32 weeks
  BMC(g) will be assessed for whole body, proximal femur on the non-dominant side (femoral nech, trochanter, intertrochanter, Ward's triangle and total hip) and lumbar spine segments (L1-L4) (L2-L4) (L1-L3) and single vertebrae (L1, L2, L3, L4) will be assessed using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change T-Score | Baseline, 16 and 32 weeks
  T-Score (SD) will be assessed for whole body, proximal femur on the non-dominant side (femoral nech, trochanter, intertrochanter, Ward's triangle and total hip) and lumbar spine segments (L1-L4) (L2-L4) (L1-L3) and single vertebrae (L1, L2, L3, L4) will be assessed using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change in Z-Score | Baseline, 16 and 32 weeks
  Z-Score (SD) will be assessed for whole body, proximal femur on the non-dominant side (femoral nech, trochanter, intertrochanter, Ward's triangle and total hip) and lumbar spine segments (L1-L4) (L2-L4) (L1-L3) and single vertebrae (L1, L2, L3, L4) will be assessed using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA)
Change in fracture risk | Baseline, 16 and 32 weeks
  Will be assessed via the FRAX ® tool.
Change in self-reported quality of life | Baseline, 16 and 32 weeks
  Will be assessed via Short form quality of life questionnaire (SF36)
Change in basic activities of daily living | Baseline
  Will be assessed via Barthel index of activities of daily living.
Change in instrumental activities of daily living | Baseline
  Will be assessed via Lawton and Brody instrumental activities of daily living scale. There are eight domains of function measured with the Lawton and Brody scale. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent).
Level of physical activity | Baseline
  The level of physical activity of the participants will be assessed by Global Physical Activity Questionnaire (GPAQ)
Cognitive function | Baseline
  The cognitive function will be assessed by the Mini Mental State Examination (MMSE) questionnaire.
Attendance to training sessions | Baseline, 16 and 32 weeks
  Daily training session attendance records will be collected by the instructors.
Adherence to training program | Week 32
  Adherence levels will be calculated at the end of the training period. Nonadherence is define as "those not attending at follow-up and have not attend for 4 weeks during the training period, and have not given a reason for nonattendance or those who have stated they are dropping out."
Change in blood pressure | Baseline, 16 and 32 weeks
  Systolic and diastolic blood pressure will be measured
Change balance based on body center of pressure | Baseline, 16 and 32 weeks
  Balance will be measured through stabilometry over different surfaces (stable or unstable) and conditions (eyes open or close)
Change in body composition-Total mass, fat-free mass and fat mass | Baseline, 16 and 32 weeks
  Total mass (Kg), fat-free mass (kg) and fat mass (kg) will be assessed for whole body and appendicular/visceral regions using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change in body composition- Percentage of body mass | Baseline, 16 and 32 weeks
  Percentage of fat mass (%) of will be assessed for whole body and appendicular/visceral regions using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change in Body mass index | Baseline, 16 and 32 weeks
  Body mass index was calculated.
Muscle quality of lower limbs | Baseline, 16 and 32 weeks
  For lower limbs will be calculated based on ratio isocinetic torque in N-m Knee flexion or extension/leg muscle mass (N-m/kg)
Muscle quality of upper limbs | Baseline, 16 and 32 weeks
  For upper limbs will be calculated based on ratio maximal grip strength arm muscle mass (Kg/Kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Physical activity and Sport Science Faculty, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No